CLINICAL TRIAL: NCT05489835
Title: Work-Health-Life-Balance 4.0 - Mental Resilience, Stability & Healthy Nutrition in a New Work Reality
Brief Title: Work-Health-Life-Balance - Mental Resilience, Stability & Healthy Nutrition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Baranyi, Assoc. Prof. Dr., Medical University of Graz
Other Study IDs: EK 34-147 ex 21/22
Record Dates: First submitted 2022-06-29; First posted 2022-08-05 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Psychological Stress; Nutritional Quality; Burn-out Syndrome; Sleep; Depressive Disorder
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological; Depressive Disorder | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employees: Employees in Austrian companies affected by digitalization
  Interventions: Behavioral: Nutritional counseling

INTERVENTIONS:
Behavioral: Nutritional counseling — Nutritional counseling

SUMMARY:
New working environments (digitalization, flexibilization) can lead to increased levels of stress. A balanced work-life balance is therefore important in order to prevent negative effects of stress on mental health.

This study investigates,

1. how stress, recovery, nutritional behavior, resilience and sleep behavior are related to the changed working conditions.
2. how standardized nutritional training affects individual body composition (measured using Bioelectrical Impedance Analyses, BIA), stress perception, burn-out symptoms and sleep.

DETAILED DESCRIPTION:
The ways of working must adapt to the challenges and opportunities of the digital world. Work 4.0 describes the process of change in the working environment in the digital age. Adapting to rapidly changing and sometimes uncertain living and working conditions in times of digitization, dislocated working (including "home office") and altered work processes demands a considerable effort of resources from numerous employees. Previously established work environments and behaviors are being evaluated and adapted to the new circumstances and requirements.

Such times of change often cause uncertainty and result in increased stress levels. Stress, in turn, leads to a variety of symptoms in many areas of life and work, which can limit the ability to work. As a result, successful adaptation to the challenges of the new work reality of Work 4.0 can fail.

Research Questions:

This study investigates,

1. how stress, recovery, nutritional behavior, resilience and sleep behavior are related to the changed working conditions and central characteristics of work 4.0.
2. how standardized nutritional training based on the Austrian Food Pyramid affects individual body composition (measured using Bioelectrical Impedance Analyses, BIA), stress perception, burn-out symptoms and sleep.

ELIGIBILITY:
Inclusion Criteria:

* employees in austrian companies affected by digitalization
* Informed consent

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: employees in austrian companies affected by digitalization
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-11 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Stress | 3 months
  Stress-Erholungsfragebogen (RESTQ); minimum value: 0, maximum value: 294; High scores reflect high subjective stress.

SECONDARY OUTCOMES:
Sleep | 3 months
  Insomnis severity index: minimum value: 0, maximum value: 28; High scores reflect the presence of sleeping disorders
Body mass index | 3 months
  Body mass index (BMI); BMI= body weight / (body height)²

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baranyi, M.D., Principal Investigator — Medical University of Graz, Auenbruggerplatz 31, 8036 Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No